CLINICAL TRIAL: NCT01198899
Title: Belgian Screening Project for the Detection of Anderson-Fabry Disease in Hypertrophic Cardiomyopathy
Status: Completed | Type: Observational
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: 2009/035
Record Dates: First submitted 2010-08-31; First posted 2010-09-10 (Estimated); Last update posted 2012-01-12 (Estimated); Status verified 2012-01

CONDITIONS: Left Ventricular Hypertrophy
Keywords: Fabry-Anderson disease; gen mutation; left ventricular hypertrophy
MeSH Terms: conditions — Hypertrophy, Left Ventricular; Fabry Disease | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- left ventricular hypertrophy: Patients with left ventricular hypertrophy will be used.
  Interventions: Other: blood sampling

INTERVENTIONS:
Other: blood sampling — Blood sampling will be used.

SUMMARY:
The purpose of this study is to determine the prevalence of Fabry mutations in patients with left ventricular hypertrophy (moderate to severe), as measured by echocardiography.This study is a screening study

ELIGIBILITY:
Inclusion Criteria:

* All patients over 18 years undergoing a routine echocardiography in the participating hospitals
* Both genders will be considered.
* Patients can be included if on 2D echocardiography the maximal septal wall thickness > 13 mm and/or the posterior wall thickness > 13 mm. The limit for inclusion is kept relatively low to detect early forms of Fabry cardiomyopathy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with left ventricular hypertrophy
Sampling Method: Non-Probability Sample
Enrollment: 540 (Actual)
Dates: Start 2009-07; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Determination of the prevalence of Fabry mutations in patients with left ventricular hypertrophy (moderate to severe), as measured by echocardiography | At baseline T0
  patients with left ventricular hypertrophy will be screened for Fabry mutations, and results will be communicated within four months

CONTACTS AND LOCATIONS:
Overall Officials: Raymond Vanholder, MD, PhD, Principal Investigator — University Hospital Ghent, Belgium
Locations (9):
- Belgium (9):
  - AZ Imelda, Bonheiden
  - AZ Sint-Blasius, Dendermonde
  - AZ Sint-Lucas, Ghent
  - Maria Middelares, Ghent
  - University Hospital Ghent, Ghent
  - Jan Yperman Ziekenhuis, Ieper
  - AZ Oostkust, Knokke-Heist
  - ZOL, Limbourg
  - AZ Zusters van Barmhartigheid, Ronse

REFERENCES:
- [Derived] Terryn W, Deschoenmakere G, De Keyser J, Meersseman W, Van Biesen W, Wuyts B, Hemelsoet D, Pascale H, De Backer J, De Paepe A, Poppe B, Vanholder R. Prevalence of Fabry disease in a predominantly hypertensive population with left ventricular hypertrophy. Int J Cardiol. 2013 Sep 10;167(6):2555-60. doi: 10.1016/j.ijcard.2012.06.069. Epub 2012 Jul 16. PMID 22805550
- See also: website of University Hospital Ghent, Belgium — http://www.uzgent.be